CLINICAL TRIAL: NCT02515838
Title: A Multi-Centre, Phase II, Randomized, Double-Blind, Placebo-Controlled Study to Investigate Efficacy and Safety of Sevuparin Infusion for the Management of Acute Vaso-Occlusive Crisis (VOC) in Subjects With Sickle-Cell Disease (SCD).
Brief Title: Sevuparin Infusion for the Management of Acute VOC in Subjects With SCD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Modus Therapeutics AB (Industry)
Collaborators: Ergomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TVOC01
Record Dates: First submitted 2015-07-27; First posted 2015-08-05 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-02

CONDITIONS: Sickle-Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — sevuparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo infusion
  Interventions: Other: Placebo
- Sevuparin (Experimental): Sevuparin infusion
  Interventions: Drug: Sevuparin

INTERVENTIONS:
Drug: Sevuparin — The Drug Product sevuparin solution for IV infusion
  Arms: Sevuparin
Other: Placebo — Placebo for IV infusion
  Arms: Placebo

SUMMARY:
A Multi-Centre, Phase II, Randomized, Double-Blind, Placebo-Controlled Study to investigate Efficacy and Safety of Sevuparin Infusion for the Management of Acute Vaso-Occlusive Crisis (VOC) in Subjects with Sickle-Cell Disease (SCD).

DETAILED DESCRIPTION:
This will be a phase II, multi-centre, randomized, double-blind, placebo-controlled study designed to assess preliminary efficacy, safety and pharmacokinetics (PK) of 2-7 days continuous IV administration of sevuparin for the management of acute VOC in subjects with SCD.

Adults and adolescents ≥ 12 years of age will be randomized to treatment with sevuparin or placebo (ratio 1:1).

ELIGIBILITY:
Inclusion Criteria:

* Sign a written informed consent (adults, parents) and assent (adolescents)
* Male or female, age 12-50 years.
* Diagnosis of Sickle cell disease
* Subjects admitted for an acute, painful VOC to be treated/or treated with parenteral opioid analgesia.
* Expectancy of need for hospitalization during at least 48 hours.
* Be at least 1 year postmenopausal, surgically sterile, or if Women of Child Bearing Potential (WOCBP), e.g. following menarche practicing an effective method of birth control

Exclusion Criteria:

* Severe hepatic failure/disease, abnormal liver enzyme tests or history of hepatitis B virus (HBV), hepatitis C virus (HCV)
* Abnormal conjugated (direct) bilirubin 3 fold above ULN
* History of clinically significant bleeding in vital organs
* Current clinically significant bleeding, as judged by the investigator
* Current use of acetylsalicylic acid (ASA), anti-platelet therapy, anticoagulant therapy
* Abnormal coagulation laboratory values
* A platelet count <75,000/µL.
* BMI >35
* Subjects with more than 5 hospitalizations for VOC during the last 6 months
* Evidence of acute SCD complications other than VOC at screening
* The use of strong opioids for > 3 consecutive days during the last 15 days before presenting to the hospital
* History of chronic drug abuse.
* Renal dysfunction
* Known infection (positivity) with human immunodeficiency virus (HIV), HBV or HCV.
* Significant ECG abnormality
* History of a clinically significant drug allergy to heparin, LMWH's, sevuparin, or morphine.
* Use of any investigational agent during the 30 days prior to the first dose.
* For females: pregnancy, lactating or intention of becoming pregnant
* Evidence of clinically significant disorders that might interfere with the study aim or safety of the subject
* Any condition that, in the view of the Investigator, places the subject at high risk of poor treatment compliance or of not completing the study.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 147 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Time to resolution of VOC | From hospitalisation until discharge, defined as freedom from parenteral opioid use and readiness for discharge i.e. from randomisation until day 7
  Time from start of infusion until resolution of VOC crisis/episode

SECONDARY OUTCOMES:
Frequency and pattern of treatment-emergent adverse event (TEAEs) | Time from start randomsiation until end of study, approximately 1 month 1 week after randomisation
  All events to be reported from randomization until end of study
Pharmacokinetic (PK) characteristics of sevuparin | Pre dose, 1h, 2h, 24h, 1/day (day 3-8)
  PK characteristics of sevuparin during and after administration of sevuparin as a continuous IV infusion (subgroup) ◦Area under the plasma concentration versus time curve (AUC) of Sevuparin.
Mean change in pain intensity | From baseline (visit 1) until day 3-7
  VAS (visual analog scale) every fourth hour. Range from 0 (no pain) to 100 (max pain)
Duration of severest pain, | From baseline (visit 1) until day 3-7
  Defined as time to a 30% reduction in pain intensity (VAS)
Cumulative dose of parenteral opioids | From baseline (visit 1) until day 3-7
  Total dose of parenteral opioids

CONTACTS AND LOCATIONS:
Overall Officials: Dr Bart J Biemond, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (20):
- Bahrain (2):
  - Salmaniya Hospital, Kingdom of Bahrain, Manama
  - Salmaniya Medical Complex, Bahrain, Manama
- Jamaica (7):
  - Annotto Bay Hospital, Annotto Bay
  - Kingston Public Hospital, Kingston
  - University Hospital of the West Indies, Kingston
  - Winchester Surgical and Medical Institute, Kingston
  - Mandeville Regional Hospital, Mandeville
  - May Pen Public Hospital Clarendon, May Pen
  - Cornwall Regional Hospital, Jamaica, Montego Bay
- Lebanon (2):
  - American University of Beirut Medical Center, Beirut, Cairo street, Beirut, Lebanon, Beirut
  - Nini Hospital, Tripoli
- Netherlands (2):
  - Dept of Haematology, Amsterdam
  - Erasmus MC, Rotterdam
- Oman (2):
  - Sultan Qaboos University Hospital Alkhodh, Oman, Muscat
  - Sultan Qaboos University, Muscat
- Saudi Arabia (2):
  - King Fahd Medical City, As Sulimaniyah, Riyadh Saudiarabien, Riyadh
  - King Saud University, Riyadh, Saudiarabien, Riyadh
- Turkey (Türkiye) (3):
  - Mersin University Faculty of Medicine, Adana, Mersin
  - Cukurova University Faculty Of Medicine Tıp Fakültesi, Adana
  - Dr Antmen, Adana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Biemond BJ, Tombak A, Kilinc Y, Al-Khabori M, Abboud M, Nafea M, Inati A, Wali Y, Kristensen J, Kowalski J, Donnelly E, Ohd J; TVOC01 Investigators Group. Sevuparin for the treatment of acute pain crisis in patients with sickle cell disease: a multicentre, randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Haematol. 2021 May;8(5):e334-e343. doi: 10.1016/S2352-3026(21)00053-3. PMID 33894169